CLINICAL TRIAL: NCT04824196
Title: Comparison of Effects of Vestibular Visual Cues and Proprioception To Improve Postural Control in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2040 Hafsa Mustafah
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Older Adults
Keywords: Postural control; Proprioception; Vestibular; Elderly; BBS; CTSIB

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vestibular visual cues therapy (Experimental): Pelvic rolling to right and left with head movement and stop first on right side for 3 minutes. Do this exercise in front of the mirror.Anterior, posterior, left, and right rectilinear stimulation activities on a therapeutic ball. Anterior, posterior, left and right rectilinear movements were performed for five minutes
  Interventions: Other: vestibular visual cues therapy
- propriocetion therapy (Active Comparator): Alternate knee flexion-extension with extended trunk posture using both hands for support.
  Hip and knee flexion-extension with swiss ball between the back and wall.
  Hip aises lying with their back on the floor with both legs on the swiss ball. Upper limbs leaning on the floor to help with the exercises.
  then perform all exercise on gym ball
  Interventions: Other: propriocetion exercise

INTERVENTIONS:
Other: vestibular visual cues therapy — Pelvic rolling to right and left with head movement and stop first on right side for 3 minutes. Do this exercise in front of the mirrorAnterior, posterior, left, and right rectilinear stimulation activities on a therapeutic ball. Anterior, posterior, left and right rectilinear
  Arms: vestibular visual cues therapy
Other: propriocetion exercise — 1. Alternate knee flexion-extension with extended trunk posture using both hands for support.
  2. Hip and knee flexion-extension with swiss ball between the back and wall.
  3. Hip raises lying with their back on the floor with both legs on the swiss ball. Upper limbs leaning on the floor to help with the exercises. then all exercise are perfomed on gym ball
  Arms: propriocetion therapy

SUMMARY:
Background/Objective: The aim of this study was to compare the effects of vestibular visual cues and propriception to improve postural control in elderly.

DETAILED DESCRIPTION:
RCT study was conducted. Fourty four healthy elderly volunteers aged from 65 years to 75 years were assigned to a group 1 (n=22) engaging in vestibular visual cues exercises and group 2 (n=22) engaging in proprioception exercises. Training sessions (~30 minutes each) occurred twice a week for consecutive six weeks. The following parameters were analyzed before and after training for both groups: Berg balance scale (BBS) and Clinical test of sensory organization and balance (CTSIB).

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk without any device or need of continuous physical assistance to support body weight or maintain balance.
* Able to follow simple directions, for example, left, right, up, or down.
* Either using visual aids.
* Fakuda test for screening.
* VOR reflex for screening

Exclusion Criteria:

* • Presence of orthopedic problems.

  * Neurological disorders.
  * Psychological problems.
  * Cognitive issues.
  * People with severe visual issues
  * Participants with other medical complications.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 2 months
  The Berg Balance Scale (or BBS) is a widely used clinical test of a person's static and dynamic balance abilities, named after Katherine Berg, one of the developers. For functional balance tests, the BBS is generally considered to be the gold standard.[3]
  The test takes 15-20 minutes and comprises a set of 14 simple balance related tasks, ranging from standing up from a sitting position, to standing on one foot. The degree of success in achieving each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores
Clinical test of sensory organization and balance (CTSIB | 2 months
  nical Test of Sensory Interaction and Balance (CTSIB) is a tool that assesses a person's ability to use sensory inputs for balance. The original test included 6 conditions: (1) standing with eyes open on a firm surface, (2) standing with eyes closed on a firm surface, (3) standing with a visual conflict dome on a firm surface, (4)

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Binash afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martins E Silva DC, Bastos VH, de Oliveira Sanchez M, Nunes MK, Orsini M, Ribeiro P, Velasques B, Teixeira SS. Effects of vestibular rehabilitation in the elderly: a systematic review. Aging Clin Exp Res. 2016 Aug;28(4):599-606. doi: 10.1007/s40520-015-0479-0. Epub 2015 Oct 28. PMID 26511625
- [Background] Kleffelgaard I, Soberg HL, Tamber AL, Bruusgaard KA, Pripp AH, Sandhaug M, Langhammer B. The effects of vestibular rehabilitation on dizziness and balance problems in patients after traumatic brain injury: a randomized controlled trial. Clin Rehabil. 2019 Jan;33(1):74-84. doi: 10.1177/0269215518791274. Epub 2018 Jul 30. PMID 30056743
- [Background] Ribeiro KM, Freitas RV, Ferreira LM, Deshpande N, Guerra RO. Effects of balance Vestibular Rehabilitation Therapy in elderly with Benign Paroxysmal Positional Vertigo: a randomized controlled trial. Disabil Rehabil. 2017 Jun;39(12):1198-1206. doi: 10.1080/09638288.2016.1190870. Epub 2016 Jun 24. PMID 27340939
- [Background] Rossi-Izquierdo M, Gayoso-Diz P, Santos-Perez S, Del-Rio-Valeiras M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Lirola-Delgado A, Soto-Varela A. Vestibular rehabilitation in elderly patients with postural instability: reducing the number of falls-a randomized clinical trial. Aging Clin Exp Res. 2018 Nov;30(11):1353-1361. doi: 10.1007/s40520-018-1003-0. Epub 2018 Jul 14. PMID 30008159
- [Background] Ricci NA, Aratani MC, Caovilla HH, Gananca FF. Effects of Vestibular Rehabilitation on Balance Control in Older People with Chronic Dizziness: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2016 Apr;95(4):256-69. doi: 10.1097/PHM.0000000000000370. PMID 26368833
- [Background] Tramontano M, Martino Cinnera A, Manzari L, Tozzi FF, Caltagirone C, Morone G, Pompa A, Grasso MG. Vestibular rehabilitation has positive effects on balance, fatigue and activities of daily living in highly disabled multiple sclerosis people: A preliminary randomized controlled trial. Restor Neurol Neurosci. 2018;36(6):709-718. doi: 10.3233/RNN-180850. PMID 30412513
- [Background] Hebert JR, Corboy JR, Manago MM, Schenkman M. Effects of vestibular rehabilitation on multiple sclerosis-related fatigue and upright postural control: a randomized controlled trial. Phys Ther. 2011 Aug;91(8):1166-83. doi: 10.2522/ptj.20100399. Epub 2011 Jun 16. PMID 21680771
- [Background] Jahn K. The Aging Vestibular System: Dizziness and Imbalance in the Elderly. Adv Otorhinolaryngol. 2019;82:143-149. doi: 10.1159/000490283. Epub 2019 Jan 15. PMID 30947233
- [Background] Eibling D. Balance Disorders in Older Adults. Clin Geriatr Med. 2018 May;34(2):175-181. doi: 10.1016/j.cger.2018.01.002. Epub 2018 Feb 24. PMID 29661330
- [Background] Melo RS, Lemos A, Paiva GS, Ithamar L, Lima MC, Eickmann SH, Ferraz KM, Belian RB. Vestibular rehabilitation exercises programs to improve the postural control, balance and gait of children with sensorineural hearing loss: A systematic review. Int J Pediatr Otorhinolaryngol. 2019 Dec;127:109650. doi: 10.1016/j.ijporl.2019.109650. Epub 2019 Aug 21. PMID 31466025